CLINICAL TRIAL: NCT02300623
Title: Long Term Follow-up of Patients Experiencing Structured Treatment Interruption (STI) With or Without Low Doses of Interleukin-2 During Primary HIV Infection (PHI)
Brief Title: Intermittent ART in Primary HIV Infection
Acronym: PHI-IL2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHI-IL2
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: HIV
MeSH Terms: interventions — Interleukin-2; Stavudine; Lamivudine; Indinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Antiretroviral therapy alone
  Interventions: Drug: Antiretroviral therapy alone
- Treatment (Experimental): Antiretroviral therapy plus Interleukin-2'
  Interventions: Drug: Antiretroviral therapy plus Interleukin-2

INTERVENTIONS:
Drug: Antiretroviral therapy plus Interleukin-2 — Daily s.c. IL-2: 750,000 UI/m2/day for 6 months
  Other Names: IL-2; Stavudine; Lamivudine; Indinavir
  Arms: Treatment
Drug: Antiretroviral therapy alone — Standard antiretroviral therapy
  Other Names: stavudine; Lamivudine; Indinavir
  Arms: Control

SUMMARY:
Interventions during primary HIV infection (PHI) can modify the immune control and the clinical evolution during the chronic phase. Although several studies suggest the benefit of antiretroviral treatment (ART) during PHI, indication of ART is still not universally recommended. The investigators randomized patients with PHI, with a favourable immunological profile and well controlled on ART, to undergone structured treatment interruptions alone or with low doses of IL-2, stopping ART thereafter. The endpoints were immune control of HIV replication and time to resume ART. Immunological profile, specific CD4 and CD8 responses and clinical data were analysed for both groups up to 48 weeks, and during a long follow-up, up to nine years since final ART stop.

DETAILED DESCRIPTION:
The study design included two phases. The first phase consisted in four STI of 8 weeks each (off-ART), separated by 16 weeks of treatment -or the time necessary to reach again to PVL <20 copies/mL- (on-ART). At the end of the 4th off-ART cycle (week 0) an interim evaluation was performed and the second phase initiated. During the second phase, the first 6 patients received ART until they reach PVL<20 copies/mL, discontinuing thereafter (final stop). The last 6 patients received ART and low doses of IL-2. ARV therapy was stopped after reaching PVL<20 copies/mL (final stop) and IL-2 after 6 months of treatment. IL-2 was prescribed at a dose of 750.000 UI/m2 daily and was self-administrated in all patients previous trained by a specialized nurse. ART was resumed in patient dropping CD4 cell count less than 350 cell/mm3 in two consecutive determinations or in patients who developed opportunistic infections. A long term follow up analysis was performed at 3, 6 and 9 years since the final stop. It included time to resume ART, clinical events, survival rate, CD4-CD8-CD4/CD8 ratio.

ELIGIBILITY:
Inclusion Criteria:

* PHI defined by detectable plasma viral load (PVL) or p24 antigen detection coupled with a negative or indeterminate LIA assay (according CDC criteria); negative HIV-1 EIA in the preceding 90 days or by a positive EIA and LIA assay with acute retroviral syndrome in the preceding 90 days of starting ART plus documented negative HIV-1 EIA within the previous year.
* ART started within 90 days from the HIV exposure and continuing in the same treatment at least 12 months before the inclusion, and they must have shown good virological and immunological responses, defined as undetectable PVL (<20 copies/mL in the last two controls) and CD4 more than 500 cells/mm3 with a CD4/CD8 ratio >1 in the last 8 months previous to enrolment

Exclusion Criteria:

* Infection of more than 90 days.
* Age under 18 years old.
* AIDS defining condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Control of viral replication without ART. | 48 weeks

SECONDARY OUTCOMES:
Time to resume ART. | 9 years after final stop

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Miró, MDPhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Sued O, Ambrosioni J, Nicolas D, Manzardo C, Aguero F, Claramonte X, Plana M, Tuset M, Pumarola T, Gallart T, Gatell JM, Miro JM. Structured Treatment Interruptions and Low Doses of IL-2 in Patients with Primary HIV Infection. Inflammatory, Virological and Immunological Outcomes. PLoS One. 2015 Jul 17;10(7):e0131651. doi: 10.1371/journal.pone.0131651. eCollection 2015. PMID 26186440